CLINICAL TRIAL: NCT03030261
Title: A Phase II Study of Elotuzumab, Pomalidomide, & Dexamethasone (Elo-Pom-Dex) With Second Autologous Stem Cell Transplantation for Relapsed Multiple Myeloma
Brief Title: Elotuzumab, Pomalidomide, & Dexamethasone (Elo-Pom-Dex) With Second Autologous Stem Cell Transplantation for Relapsed Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Bristol-Myers Squibb (Industry); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201701084; CA204-225 (Other: Bristol-Myers Squibb); PO-CL-MM-PI-008341 (Other: Celgene)
Record Dates: First submitted 2017-01-18; First posted 2017-01-24 (Estimated); Results first posted 2023-12-15 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma in Relapse
MeSH Terms: interventions — elotuzumab; pomalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Elotuzumab + Pomalidomide + Dexamethasone (Experimental): * Patients will receive 2-6 cycles of salvage/induction per standard of care. After protocol version 02/13/2020, patients may have already received their induction therapy prior to enrolling in the study.
  * Following induction, patients will undergo standard of care ASCT melphalan conditioning (ASCT). Administration of melphalan and the second ASCT will be done as part of routine care and procedures are not dictated by this protocol.
  * Continuation therapy with Elo-Pom-Dex will begin between Days 80 and 120 following the second ASCT:
    * 10 mg/kg of elotuzumab on Days 1 and 15 for Cycles 1-6 followed by 20 mg/kg on Day 1 for Cycles 7+
    * 2 mg pomalidomide daily on Days 1-21 of all cycles
    * 40 mg dexamethasone on Days 1 and 15 of all cycles for Cycles 1-6 followed by 40 mg on Day 1 for Cycles 7+
  * Continuation therapy may continue until relapse or progression.
  Interventions: Drug: Elotuzumab; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Elotuzumab — During continuation therapy, elotuzumab will be administered on a 28-day cycle as follows: on Days 1 and 15 for Cycles 1-6 and on Day 1 for Cycles 7+. For Cycles 1-6 elotuzumab will be administered intravenously at a dose of 10 mg/kg. For Cycles 7+ elotuzumab will be administered at a dose of 20 mg/kg.
  Other Names: Empliciti
Drug: Pomalidomide — During continuation therapy, pomalidomide will be taken by mouth daily on Days 1-21 of each 28-day cycle at a starting dose of 2 mg. During continuation, pomalidomide may be dose escalated to 4 mg at the discretion of the treating physician if the 2 mg dose is tolerated.
  Other Names: Pomalyst
Drug: Dexamethasone — During continuation therapy, dexamethasone will be taken by mouth at a starting dose of 40 mg. It will be given on a 28-day cycle as follows: on Days 1 and 15 for Cycles 1-6 and on Day 1 only for Cycles 7+. Sufficient quantity of drug for one cycle of therapy will be prescribed to the patient at a time.
  Other Names: Decadron

SUMMARY:
Based on the need to improve outcomes post second autologous stem cell transplant (ASCT) for multiple myeloma (MM) and the benefits seen of maintenance treatment following initial ASCT, the natural next step is to evaluate maintenance/continuation therapy following second ASCT.

Pomalidomide is active against MM cells refractory to both bortezomib and lenalidomide, making it an ideal choice for continuation therapy following second ASCT. Adding elotuzumab may increase efficacy and also the durability of responses which is essential to improving outcomes following second ASCT.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of multiple myeloma.
* Received prior autologous stem cell transplantation as first line therapy for multiple myeloma with subsequent disease relapse/progression.
* Failed 1 or 2 lines of treatment for multiple myeloma. A line of treatment includes all therapy including induction, transplant, and maintenance administered in a sequence in the absence of relapse/progression. Once relapse/progression occurs and subsequently the anti-myeloma treatment is changed, a new line of treatment has begun. Local radiation or corticosteroids will not be considered treatment for multiple myeloma.
* Received 2 to 6 cycles of induction therapy per standard of care prior to 2nd autologous stem cell transplantation
* Received standard of care melphalan conditioning for 2nd autologous stem cell transplantation, is currently Day +80 to +120 following transplant, and is responding to therapy (partial response or better as compared to pre-induction assessment.
* All US study participants must be registered into the mandatory POMALYST REMS® program and be willing and able to comply with the requirements of the POMALYST REMS® program. For Canadian sites, patients will followed according to the Pomalidomide pregnancy prevention program
* Females of reproductive potential within the US must agree to adhere to the scheduled pregnancy testing as required in the POMALYST REMS® program. For Canadian sites, patients will followed according to the Pomalidomide pregnancy prevention program
* At least 18 and no more than 75 years of age at enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Normal bone marrow and organ function as defined as ALL of the following:

  * Absolute neutrophil count ≥ 1000/mm^3
  * Platelets ≥ 75,000/mm^3 (transfusions not permitted within 7 days of screening)
  * Total bilirubin ≤ 2.0 x institutional upper limit of normal (IULN)
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine clearance ≥ 15 mL/min
* Females of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry through Day +100 visit. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an Institutional Review Board (IRB) approved written informed consent document.

Exclusion Criteria:

* Refractory to elotuzumab and/or pomalidomide, defined as progressive disease or clinical relapse on therapy or within 60 days following completion of therapy. Prior exposure to elotuzumab and/or pomalidomide is allowed as long as patient is not refractory to these agents.
* More than one prior transplant prior to study entry with the exception of tandem transplantation. Tandem transplantation is defined as two autologous stem cell transplants that occur within 9 months of one another, and the patient did not have disease progression in the period between the two transplants.
* Presence of peripheral neuropathy ≥ grade 3 based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v 4.0
* History of plasma cell leukemia or MM central nervous system (CNS) involvement.
* Receiving renal replacement therapy, hemodialysis, or peritoneal dialysis.
* Diagnosed with another concurrent malignancy requiring treatment.
* Known HIV or active hepatitis A, B, or C. Antidoby testing not required for screening
* Known hypersensitivity to pomalidomide, dexamethasone, or any excipients in elotuzumab, formulation, or recombinant protein
* Receiving any other investigational agents within 14 days prior to enrollment.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Females of childbearing potential must have two negative pregnancy tests. The first test should be performed within 10-14 days of study entry, and the second test within 24 hours prior to prescribing pomalidomide.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2027-09-26 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Vij, M.D., Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (2):
  - Colorado Blood Cancer Institute (Sarah Cannon), Denver, Colorado
  - Washington University School of Medicine, St Louis, Missouri
- University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Elotuzumab + Pomalidomide + Dexamethasone
Started | 25
Completed | 20
Not Completed | 5
Not completed — Still receiving continuation therapy | 5

BASELINE CHARACTERISTICS:
Arm/Group | Elotuzumab + Pomalidomide + Dexamethasone
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 62 [46 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 9
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS) Rate
Description: -Event-free survival (EFS) will be defined as time from ASCT to disease progression, relapse, or death, whichever occurs first. Patients who are removed from study therapy prior to any of these events occurring will be censored at the time of initiation of subsequent anti-myeloma treatment.
Time Frame: 1 year
Population: Only 18 patients were evaluable for this outcome measure. 6 patients did not have ASCT and 1 patient had ASCT but did not start continuation treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Elotuzumab + Pomalidomide + Dexamethasone
Number analyzed (Participants) | 18
Participants | 13

2. Secondary Outcome: Overall Response Rate (ORR)
Description: -Overall response rate (ORR) will be defined as the proportion of evaluable patients meeting the criteria for partial response (PR), very good partial response (VGPR), complete response (CR), or stringent complete response (sCR).
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Elotuzumab + Pomalidomide + Dexamethasone
Number analyzed (Participants) | 18
Participants | 18

3. Secondary Outcome: Complete Response Rate (CRR)
Description: * Complete response rate (CRR) will be defined as the proportion of evaluable patients meeting the criteria complete (CR) or stringent complete response (sCR)
  * Stringent complete response (sCR) requires all of the following:
    * CR as defined below
    * Normal free light chain ratio (0.26-1.65)
    * Absence of clonal cells in the bone marrow by immunohistochemistry or immunofluorescence
  * Complete response (CR) requires all of the following:
    * Disappearance of monoclonal protein by both protein electrophoresis and immunofixation studies from the blood and urine
    * If serum and urine monoclonal protein are unmeasurable, Normal free light chain ratio (0.26-1.65)
    * <5% plasma cells in the bone marrow
    * Disappearance of soft tissue plasmacytoma
  * Patients who do not meet the definition of CR based solely on residual monoclonal protein on serum electrophoresis and/or immunofixation, but are MRD-negative as described above, will also be considered CR.
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Elotuzumab + Pomalidomide + Dexamethasone
Number analyzed (Participants) | 18
Participants | 12

4. Secondary Outcome: Progression-free Survival (PFS)
Description: -Progression-free survival (PFS) will be defined as time from ASCT to disease progression or relapse. Any patient who expires or withdraws prior to disease progression or relapse will be censored at last follow-up. Patients who are removed from study therapy prior to progression or relapse will be censored at the time of initiation of subsequent anti-myeloma treatment.
Time Frame: Up to 5 years post completion of treatment
Reporting Status: Not Posted

5. Secondary Outcome: Overall Survival (OS)
Description: -Overall survival (OS) will be defined as time from ASCT to death due to any causes. Patients who are alive at the time of data analyses will be censored on the last known alive date. Patients who are removed from study therapy prior death will be censored at the time of initiation of subsequent anti-myeloma treatment.
Time Frame: Up to 5 years post completion of treatment
Reporting Status: Not Posted

6. Secondary Outcome: Toxicity of Regimen as Measured by Number of Grade 3-5 Adverse Events
Description: -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Time Frame: Up to 30 days following completion of treatment (estimated to be 106 weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: -Following induction and continuation therapy, AEs & all-cause mortality are collected from start of treatment through 30 days after treatment completion or the start of next anti-myeloma therapy. AEs were followed for median of 434 days, full range 83-1424 days. -During the follow-up phase, all-cause mortality data are collected through 5 years after treatment completion, up to 10 years. All-cause mortality were followed for median of 884 days, full range 187-1948 days.
Description: The follow-up group is to show all-cause mortality only. Induction On Study group will show AEs and SAEs that occurred during that treatment time period and 30 days after that treatment time period if they stopped treatment in that time period. The Continuation group will show AEs and SAE that occurred during that treatment time period and for 30 days after that treatment time period if they stopped treatment in that time period.
Groups:
- Induction Therapy On Study: -Patients will receive 2-6 cycles of salvage/induction per standard of care. After protocol version 02/13/2020, patients may have already received their induction therapy prior to enrolling in the study.
- Continuation: * Continuation therapy with Elo-Pom-Dex will begin between Days 80 and 120 following the second ASCT:
    * 10 mg/kg of elotuzumab on Days 1 and 15 for Cycles 1-6 followed by 20 mg/kg on Day 1 for Cycles 7+
    * 2 mg pomalidomide daily on Days 1-21 of all cycles
    * 40 mg dexamethasone on Days 1 and 15 of all cycles for Cycles 1-6 followed by 40 mg on Day 1 for Cycles 7+
  * Continuation therapy may continue until relapse or progression.
- Follow-up: -Participants will be followed annually for up to 5 years after removal from study or until death, whichever occurs first.
Arm/Group | Induction Therapy On Study | Continuation | Follow-up
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18 | 8/25
Serious Adverse Events (participants affected / at risk) | 6/16 | 7/18 | 0/0
Other Adverse Events (participants affected / at risk) | 16/16 | 18/18 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Therapy On Study (N=16) | Continuation (N=18) | Follow-up (N=0)
Heart failure (Cardiac disorders) | 0 | 0 | NA
Myocardial infarction (Cardiac disorders) | 0 | 1 | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | NA
Diarrhea (Gastrointestinal disorders) | 1 | 1 | NA
Fatigue (General disorders) | 0 | 0 | NA
Fever (General disorders) | 0 | 0 | NA
Infusion related reaction (General disorders) | 0 | 1 | NA
E. coli sepsis (Infections and infestations) | 0 | 1 | NA
Lung infection (Infections and infestations) | 2 | 2 | NA
Rhinovirus (Infections and infestations) | 0 | 1 | NA
Sepsis (Infections and infestations) | 0 | 1 | NA
Staph lugdunensis right toe (Infections and infestations) | 0 | 1 | NA
Upper respiratory infection (Infections and infestations) | 1 | 3 | NA
Urinary tract infection (Infections and infestations) | 2 | 0 | NA
Acute kidney injury (multiple myeloma progression) (Renal and urinary disorders) | 0 | 1 | NA
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Therapy On Study (N=16) | Continuation (N=18) | Follow-up (N=0)
Anemia (Blood and lymphatic system disorders) | 8 | 3 | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | NA
Atrial fibrillation (Cardiac disorders) | 1 | 2 | NA
Chest pain (Cardiac disorders) | 2 | 1 | NA
Chest tightness (Cardiac disorders) | 0 | 0 | NA
Palpitations (Cardiac disorders) | 0 | 3 | NA
Sinus bradycardia (Cardiac disorders) | 1 | 0 | NA
Sinus tachycardia (Cardiac disorders) | 1 | 1 | NA
Earwax buildup (Ear and labyrinth disorders) | 0 | 1 | NA
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | NA
Blurred vision (Eye disorders) | 0 | 1 | NA
Double vision (Eye disorders) | 0 | 1 | NA
Dry eye (Eye disorders) | 0 | 1 | NA
Glaucoma (Eye disorders) | 0 | 1 | NA
Haze on left eye (Eye disorders) | 1 | 0 | NA
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | NA
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | NA
Constipation (Gastrointestinal disorders) | 4 | 7 | NA
Diarrhea (Gastrointestinal disorders) | 5 | 10 | NA
Dry mouth (Gastrointestinal disorders) | 0 | 2 | NA
Gastroenteritis (Gastrointestinal disorders) | 1 | 0 | NA
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | NA
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | NA
Nausea (Gastrointestinal disorders) | 5 | 6 | NA
Oral pain (Gastrointestinal disorders) | 0 | 1 | NA
Toothache (Gastrointestinal disorders) | 0 | 1 | NA
Vomiting (Gastrointestinal disorders) | 2 | 3 | NA
Chills (General disorders) | 2 | 0 | NA
Edema limbs (General disorders) | 3 | 4 | NA
Fatigue (General disorders) | 10 | 8 | NA
Fever (General disorders) | 5 | 3 | NA
Flu like symptoms (General disorders) | 1 | 2 | NA
Flushing (General disorders) | 1 | 0 | NA
IV pain (General disorders) | 0 | 1 | NA
Infusion related reaction (General disorders) | 2 | 1 | NA
Localized edema (General disorders) | 0 | 1 | NA
Malaise (General disorders) | 1 | 1 | NA
Neck edema (General disorders) | 0 | 1 | NA
Non-cardiac chest pain (General disorders) | 2 | 3 | NA
Pain (General disorders) | 3 | 0 | NA
Sweating (General disorders) | 1 | 0 | NA
CMV (Infections and infestations) | 1 | 0 | NA
CMV Bacteremia (Infections and infestations) | 0 | 1 | NA
Cellulitis - right foot (Infections and infestations) | 0 | 1 | NA
Clostridium difficile (Infections and infestations) | 0 | 1 | NA
Ear infection (Infections and infestations) | 0 | 1 | NA
Enterocolitis infectious (Infections and infestations) | 1 | 1 | NA
Fungemia (Infections and infestations) | 1 | 0 | NA
Gram negative bacteremia (Infections and infestations) | 0 | 1 | NA
Gum infection (Infections and infestations) | 1 | 0 | NA
Lip infection (Infections and infestations) | 1 | 1 | NA
Lung infection (Infections and infestations) | 1 | 5 | NA
Nail infection (Infections and infestations) | 0 | 1 | NA
Sinusitis (Infections and infestations) | 0 | 2 | NA
Upper respiratory infection (Infections and infestations) | 9 | 7 | NA
Urinary tract infection (Infections and infestations) | 0 | 2 | NA
Bruising (Injury, poisoning and procedural complications) | 1 | 2 | NA
Fall (Injury, poisoning and procedural complications) | 2 | 9 | NA
Fracture (Injury, poisoning and procedural complications) | 1 | 2 | NA
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA
Venous injury (Injury, poisoning and procedural complications) | 0 | 1 | NA
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | NA
Alanine aminotransferase increased (Investigations) | 5 | 7 | NA
Alkaline phosphatase increased (Investigations) | 4 | 3 | NA
Aspartate aminotransferase increased (Investigations) | 4 | 4 | NA
Blood bilirubin increased (Investigations) | 1 | 1 | NA
Cardiac troponin I increased (Investigations) | 1 | 0 | NA
Creatinine increased (Investigations) | 2 | 2 | NA
Lymphocyte count decreased (Investigations) | 11 | 8 | NA
Neutrophil count decreased (Investigations) | 10 | 7 | NA
Platelet count decreased (Investigations) | 9 | 5 | NA
Weight gain (Investigations) | 1 | 0 | NA
Weight loss (Investigations) | 1 | 0 | NA
White blood cell decreased (Investigations) | 9 | 6 | NA
Anorexia (Metabolism and nutrition disorders) | 0 | 3 | NA
Dehydration (Metabolism and nutrition disorders) | 3 | 3 | NA
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2 | NA
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 4 | NA
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2 | NA
Hypermagenesemia (Metabolism and nutrition disorders) | 1 | 0 | NA
Hypernatremia (Metabolism and nutrition disorders) | 2 | 2 | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 2 | NA
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 3 | NA
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | NA
Hypokalemia (Metabolism and nutrition disorders) | 4 | 4 | NA
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | NA
Hyponatremia (Metabolism and nutrition disorders) | 4 | 2 | NA
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 4 | NA
Thirst (Metabolism and nutrition disorders) | 1 | 0 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 7 | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | NA
Interscapular pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA
Jaw pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | NA
Leg and hand cramps (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA
Leg cramps (Musculoskeletal and connective tissue disorders) | 1 | 1 | NA
Leg pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA
Muscle cramping (Musculoskeletal and connective tissue disorders) | 1 | 1 | NA
Muscle spasm in back (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA
Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 5 | NA
Rib pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | NA
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | NA
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA
Amnesia (Nervous system disorders) | 1 | 0 | NA
Concentration impairment (Nervous system disorders) | 0 | 1 | NA
Dizziness (Nervous system disorders) | 8 | 5 | NA
Dysgeusia (Nervous system disorders) | 0 | 1 | NA
Encephalopathy (Nervous system disorders) | 0 | 1 | NA
Headache (Nervous system disorders) | 3 | 6 | NA
Paresthesia (Nervous system disorders) | 1 | 1 | NA
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1 | NA
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 2 | NA
Presyncope (Nervous system disorders) | 0 | 2 | NA
Syncope (Nervous system disorders) | 0 | 1 | NA
Transient ischemic attacks (Nervous system disorders) | 1 | 0 | NA
Anxiety (Psychiatric disorders) | 1 | 0 | NA
Confusion (Psychiatric disorders) | 1 | 0 | NA
Depression (Psychiatric disorders) | 1 | 0 | NA
Insomnia (Psychiatric disorders) | 3 | 2 | NA
Mood changes on dexamethasone days (Psychiatric disorders) | 1 | 1 | NA
Restlessness (Psychiatric disorders) | 1 | 0 | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | NA
Hematuria (Renal and urinary disorders) | 1 | 1 | NA
Proteinuria (Renal and urinary disorders) | 2 | 0 | NA
Urinary frequency (Renal and urinary disorders) | 0 | 1 | NA
Urinary pressure post void (Renal and urinary disorders) | 0 | 1 | NA
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | NA
Urinary tract pain (Renal and urinary disorders) | 0 | 2 | NA
Urinary urgency (Renal and urinary disorders) | 0 | 1 | NA
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 10 | NA
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA
Post nasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA
Runny nose (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | NA
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | NA
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | NA
Foot callus (Skin and subcutaneous tissue disorders) | 0 | 1 | NA
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 4 | NA
Open lesions to right and left ear (Skin and subcutaneous tissue disorders) | 0 | 1 | NA
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | NA
Purdigo nodularis (Skin and subcutaneous tissue disorders) | 0 | 1 | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | NA
Red spot under chin (Skin and subcutaneous tissue disorders) | 1 | 0 | NA
Squamous cell carcinoma (Skin and subcutaneous tissue disorders) | 0 | 1 | NA
Hematoma (Vascular disorders) | 2 | 1 | NA
Hot flashes (Vascular disorders) | 3 | 0 | NA
Hypertension (Vascular disorders) | 3 | 2 | NA
Hypotension (Vascular disorders) | 2 | 4 | NA
Peripheral vascular disease (Vascular disorders) | 0 | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/61/NCT03030261/Prot_SAP_000.pdf